CLINICAL TRIAL: NCT06331533
Title: Effects of Botulinum Toxin Type a Treatment on Clinical and Biophysical Parameters in Patients With Erythematotelangiectatic Rosacea: A Prospective, Randomized, Placebo-controlled, Double-masked Study
Brief Title: Intradermal BoNT-A Treatment in Erythematotelangiectatic Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Buğra Burç Dağtaş, Principal Investigator, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulTRH1
Record Dates: First submitted 2024-03-17; First posted 2024-03-26 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Erythematotelangiectatic Rosacea
MeSH Terms: conditions — Rosacea | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, split face, efficacy study
Who Masked: Participant, Outcomes Assessor
Masking Description: Botulinum toxin will be injected into one randomly selected half of the face, and placebo will be injected into the other half of the face. The patient will not know which half of the face was treated. An independent, blinded dermatologist will evaluate the results of the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botulinum toxin A (Experimental): 30 points were marked on a randomly selected face half at 0.5 cm intervals. 0.5 U BoNT-A was injected into each point, making a total of 15 U BoNT-A.
  Interventions: Drug: Botulinum toxin A
- Placebo (Placebo Comparator): 30 points were marked on a randomly selected face half at 0.5 cm intervals. 1.5 ml isotonic NaCl was injected intradermally into 30 points.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum toxin A — Intradermal botulinum toxin A was applied to the treatment side
  Other Names: Botox
  Arms: Botulinum toxin A
Drug: Placebo — NaCl was injected into the placebo side
  Other Names: %0.9 Sodium chloride
  Arms: Placebo

SUMMARY:
Investigation of the effectiveness of intradermal botulinum toxin A treatment in the treatment of erythematotelangiectatic rosacea (ETR) using clinical, biophysical, dermatoscopic and videocapillaroscopy.

DETAILED DESCRIPTION:
There is no gold standard treatment for erythematotelangiectatic rosacea (ETR). In recent years, some studies have been conducted to demonstrate the efficacy of intradermal botulinum toxin A (BoNT-A) treatment in ETR and facial erythema. Studies including objective and quantitative measurements are limited.

This study aims to investigate the efficacy and safety of intradermal BoNT-A treatment in ETR patients.

This randomised, double-blind, split-face study included 30 participants with erythematotelangiectatic rosacea (ETR). They were randomly randomised to intradermal BoNT-A on one side of the face and placebo on the other side. Clinician's erythema assessment (CEA) score, patient self-assessment (PSA) score, erythema index (EI), melanin index (MI), dermatoscopic and capillaroscopic analyses of background erythema and vascular structure were assessed at baseline and one month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Erythematotelangiectatic rosacea subtype
* Willingness to participate in the research and providing informed consent

Exclusion Criteria:

* Patients under 18 years of age, over 60 years of age
* A rosacea subtype other than ETR
* History of using topical or systemic medications within the past two weeks due to rosacea or other dermatoses
* Known history of autoimmune disease
* History of neuromuscular disease
* History of facial botulinum toxin injection within the last six months
* Reporting allergy to the active ingredient
* Pregnant or breastfeeding patients
* Patients who do not accept treatment and follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of erythema with Clinician's Erythema Assessment scale | One month
  The effect of intradermal BoNT-A treatment on facial erythema was evaluated using the Clinician's Erythema Assessment scale.
Evaluation of erythema using mexameter | One month
  Evaluation of the effect of intradermal BoNT-A treatment on the objective erythema value measured by mexameter.
Evaluation of erythema by dermatoscopy | One month
  Evaluation of the effect of intradermal BoNT-A treatment on dermatoscopic background erythema.

SECONDARY OUTCOMES:
Evaluation of the change in vascular structure using videocapillaroscopy | One month
  The secondary objective of the study was to examine the effect of intradermal BoNT-A treatment on the Investigator Global Assessment (poorly defined vasculature and increased vessel diameter were considered poor response; IGA score=-1, localized or complete obliteration of vascular structures was considered good; IGA score=1, no change in vascular structures was considered no response; IGA score=0) scale developed using videocapillaroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No